CLINICAL TRIAL: NCT00611819
Title: Open, Randomized and Multicenter Phase IV Study to Compare the Efficacy and Safety of Two Different Treatments Duration 24 Versus 48 Weeks in Chronic Hepatitis C Genotypes 2 and/or 3 co-Infected HIV-HCV Patients.
Brief Title: Two Different Treatments 24 vs 48 Weeks Chronic Hepatitis C Genotypes 2 and/or 3 in co-Infected HIV-HCV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Enrique Ortega, Hospital General Universitario of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHRONOS; 2005-000203-34
Record Dates: First submitted 2008-01-25; First posted 2008-02-11 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Hepatitis C; Co-Infection HIV-HCV
Keywords: hepatitis; co-infection
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Coinfection | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Peg interferon alpha 2a 180 mc/weekly Ribavirin 800 mg/daily during 24 weeks
  Interventions: Drug: Peg interferon + Ribavirin
- 2 (Active Comparator): Peg interferon alpha 2a 180 mc/weekly Ribavirin 800 mg/daily during 48 weeks
  Interventions: Drug: Peg interferon + Ribavirin

INTERVENTIONS:
Drug: Peg interferon + Ribavirin — Peg interferon 180 mcg/weekly Ribavirin 800 mg/daily during 24 weeks
  Other Names: Pegasys
  Arms: 1
Drug: Peg interferon + Ribavirin — Peg interferon alpha 2a 180 mc/weekly Ribavirin 800 mg/daily during 48 weeks
  Other Names: Pegasys
  Arms: 2

SUMMARY:
The rapidly progression of the disease in HIV-HCV co-infected patients justify the treatment.

Combination of Peg interferon and Ribavirin is the best treatment because it improve the compliance of treatment.

In APRICOT study genotypes 2 and 3 patients received 48 weeks and the rates of end of treatment response was 64% and the sustained virological response (24 weeks after the end of treatment) 62%.

In mono-infected patients trials showed there are not differences in the sustained virological response between 24 and 48 weeks of treatment, however exit the doubt concerning the different kinetic viral in HIV-HCV co-infected patients and this could be related with a lost of profit with a shorter duration of treatment, only 24 weeks.

In this study we woud like to evaluate if 24 weeks of treatment in HIV-HCV co-infected patients genotype 2 or 3 will have the same rate of clearance of virus at the end of follow-up period.

DETAILED DESCRIPTION:
Patients will randomized to receive 180 µg/weekly of Pef interferon alpha-2a and 800 mg/daily of Ribavirin during 24 weeks or 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of 18-65 years of age
* Serologic evidence of chronic hepatitis C infection by detectable plasma HCV-RNA
* Serologic evidence of HIV-1 infection by ELISA and Western-blot
* Stable status of HIV-1 infection in the opinion of the investigator
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug. Additionally, all fertile males and females must be using two forms of effective contraception during treatment and during the 6 months after treatment end. This may include, but is not limited to, using birth control pills, IUDs, condoms, diaphragms, or implants, being surgically sterilized, or being in a post-menopausal state.
* Willingness to give written informed consent and willingness to participate to and comply with the study

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* IFN or ribavirin therapy at any previous time
* Any investigational drug <6 weeks prior to the first dose of study drug
* History or other evidence of a medical condition associated with chronic liver disease other than HCV
* Hepatocarcinoma observed
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Active HIV-related opportunistic infection and/or malignancy requiring acute systemic therapy
* Absolute neutrophil count <1500 cells/mm3
* Hgb <12 g/dL in women or 13 g/dL in men or any patient for whom anemia would be medically problematic
* Hemoglobinopathy (e.g. thalassemia) or any other cause of or tendency for hemolysis
* Platelet count <90000 cells/mm3
* Serum creatinine level >1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis)
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of significant cardiac disease that could be worsened by acute anemia
* History of thyroid disease poorly controlled on prescribed medications. Patients with elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease are excluded
* Evidence of severe retinopathy
* History of major organ transplantation with an existing functional graft
* History or other evidence of severe illness, malignancy or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) <6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* Drug use within 6 months of 1st dose and excessive alcohol consumption

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
% of patients with RNA-HCV undetectable 24 weeks | 24 weeks after the end of treatment

SECONDARY OUTCOMES:
% of patients at the end of treatment | 48 weeks of treatmemt

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Ortega, Dr, Study Director — Hospital General Universitario de Valencia
Locations (18):
- Spain (18):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital de Elche, Elche, Alicante
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital General de Castellón, Castellon, Castellón
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Clínico San Cecilio, Granada, Granada
  - Hospital Infanta Elena, Huelva, Huelva
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital la Paz, Madrid, Madrid
  - Hospital General de Murcia, Murcia, Murcia
  - Hospital Carlos Haya, Málaga, Málaga
  - Hospital Xeral-Cíes, Vigo, Pontevedra
  - Hospital Virgen Macarena, Seville, Sevilla
  - Hospital de Gandia, Gandia, Valencia
  - Hospital la Fe, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia, Valencia